CLINICAL TRIAL: NCT04307732
Title: Impact of Preoperative Nutritional Status on the Postoperative Mortality and Morbidity in Patients Undergoing Valvular Heart Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-0024
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Patients Undergoing Valvular Heart Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators investigated the clinical impacts of preoperative nutritional status on mortality in patients undergoing valvular heart surgery. Preoperative nutritional status was evaluated by the prognostic nutritional index (PNI), Geriatric Nutritional Risk Index (GNRI), and controlling nutritional status (CONUT) score. The primary outcome was the association between preoperative nutritional status evaluated by PNI, GNRI, and CONUT score and postoperative mortality. The predictive discrimination ability for mortality between PNI, GNRI, and CONUT were compared. Risk factors for mortality were identified.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent valvular heart surgery from January 2013 to February 2018

Exclusion Criteria:

* Patients younger than 18 years
* Patients undergoing combined congenital heart surgery
* Patients undergoing transcatheter valve replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Terticary care hospital
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
postoperative mortality according to peroperative nutritional status | 1 year after surgery
  The association between preoperative nutritional status evaluated by the prognostic nutritional index (PNI), Geriatric Nutritional Risk Index (GNRI), and controlling nutritional status (CONUT) score and postoperative mortality is evaluated.
postoperative mortality according to peroperative nutritional status | 2 year after surgery
  The association between preoperative nutritional status evaluated by the prognostic nutritional index (PNI), Geriatric Nutritional Risk Index (GNRI), and controlling nutritional status (CONUT) score and postoperative mortality is evaluated.

SECONDARY OUTCOMES:
predictive discrimination ability for mortality between PNI, GNRI, and CONUT | 1 year after surgery
  The predictive discrimination abilities for mortality between PNI, GNRI, and CONUT score are compared.
predictive discrimination ability for mortality between PNI, GNRI, and CONUT | 2 year after surgery
  The predictive discrimination abilities for mortality between PNI, GNRI, and CONUT score are compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho JS, Shim JK, Kim KS, Lee S, Kwak YL. Impact of preoperative nutritional scores on 1-year postoperative mortality in patients undergoing valvular heart surgery. J Thorac Cardiovasc Surg. 2022 Oct;164(4):1140-1149.e3. doi: 10.1016/j.jtcvs.2020.12.099. Epub 2021 Jan 5. PMID 33551075